CLINICAL TRIAL: NCT03053999
Title: Variables That Are Correlated to Developing Multiple Endocrine Neoplasia (MEN) and Pancreatic Neuroendocrine Tumors (PNET)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA12-0892
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Multiple Endocrine Neoplasia; Pancreatic Neuroendocrine Tumors; Hyperparathyroidism
Keywords: Multiple Endocrine Neoplasia; Pancreatic Neuroendocrine Tumors; Hyperparathyroidism; HPTH; PNET; Biomarkers; Parathyroidectomy; Genome sequencing; Data review
MeSH Terms: conditions — Multiple Endocrine Neoplasia; Hyperparathyroidism; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parathyroidectomy Tissue and Data: Analyses includes genome sequencing based analysis to identify novel germline variations in blood DNAs and somatic changes in tumor DNAs, which may contribute to the development of pancreatic tumors.
  Clinical information retrieved from the patients' medical record including: de-identified demographic data (age, gender, race/ethnicity), medical history, family history, disease status, treatment response, survival information, and selected clinical data from medical record (calcium levels, calcitonin levels).
  Interventions: Other: Genome Sequencing; Other: Data Review

INTERVENTIONS:
Other: Genome Sequencing — Analyses includes genome sequencing based analysis to identify novel germline variations in blood DNAs and somatic changes in tumor DNAs, which may contribute to the development of pancreatic tumors.
Other: Data Review — Clinical information retrieved from the patients' medical record including: de-identified demographic data (age, gender, race/ethnicity), medical history, family history, disease status, treatment response, survival information, and selected clinical data from medical record (calcium levels, calcitonin levels).

SUMMARY:
The study aims to identify predictors of disease in patients with hyperparathyroidism (HPTH) who undergo surgery.

DETAILED DESCRIPTION:
Researchers aim to identify somatic mutations and inherited genetic variants which may help predict the development of PNET in patients with hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. MEN1 patients who have undergone parathyroidectomy and did not develop PNET.
2. MEN1 patients who have undergone parathyroidectomy and had surgical removal of PNET.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants identified as follows: Patients of the Surgical team at MD Anderson Cancer Center who have undergone parathyroidectomy.
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2012-10-09 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Identification of Somatic Mutations and Inherited Genetic Variants to Help Predict the Development of Pancreatic Neuroendocrine Tumors (PNET) in Participants with Hyperparathyroidism by Genome Sequencing | 10 years

SECONDARY OUTCOMES:
Identification of Somatic Mutations and Inherited Genetic Variants to Help Predict the Development of Pancreatic Neuroendocrine Tumors (PNET) in Participants with Hyperparathyroidism by Data Review | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org